CLINICAL TRIAL: NCT04106037
Title: Nosocomial and Community Acquired Legionella Pneumophila Pneumonia, a Retrospective Case Series
Brief Title: Nosocomial and Community Acquired Legionella Pneumophila Pneumonia.
Status: Completed | Type: Observational
Sponsor: Dr Philippe CLEVENBERGH (Other)
Responsible Party: Sponsor-Investigator, Dr Philippe CLEVENBERGH, Head of Infectious Diseases Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Moretti
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Legionnaires' Disease
MeSH Terms: conditions — Legionnaires' Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Legionnaires' disease: All confirmed human cases of Legionnaires' disease diagnosed within the CHU Brugmann hospital within the last 3 years: from 01/01/2016 till 31/12/2018. A similar approach will be followed for the St Pierre Hospital and the UZ Brussel Hospital.
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Legionnaire's disease (LD) is a major cause of both community acquired and nosocomial pneumonia, with Legionella pneumophila serogroup A (Lp1) being the most virulent and the greatest cause of disease. Sample culture of low respiratory tract is considered the gold standard in the diagnosis of LD, however its sensitivity seems to be poor and its performance is technically demanding. The introduction of urinary antigen detection testing (LUA) brought a major advance in LD diagnosis, with upt to 95% of cases in Europe being diagnosed with this method. Despite the high sensitivity of LUA for Lp1, ranging from 80-90%, its negative predictive value is low in other serogroup than Lp1 and therefore, Legionella may be unrecognized as agent of pneumonia. Although underdiagnosed and underreported, LD represents the second most common cause of pneumonia requiring admission in intensive care unit (ICU). Average fatality rate of LD in Europe reaches 10%, but its mortality is considered to be even higher in nosocomial patients.

Despite the higher fatality rate in hospitalized LD patients, poor is the knowledge on the risk factors that could induce disease and that increase mortality in the hospitalized population affected by LD. In order to shed more light on this topic a cohort of patients diagnosed with LD in the last 3 years will be retrospectively examined.

ELIGIBILITY:
Inclusion Criteria:

All confirmed human cases of Legionnaires' disease diagnosed within the CHU Brugmann hospital within the last 3 years, from 01/01/2016 till 31/12/2018. A similar approach will be followed for the St Pierre and the UZ Brussel Hospitals.

Exclusion Criteria:

Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All confirmed human cases of Legionnaires' disease diagnosed within the CHU Brugmann hospital, the St Pierre Hospital and the UZ Brussel Hospital. The definition of Legionnaires' disease diagnosis is met whether a seroconversion is detected or positive respiratory samples cultures are objectivized or positive LUA are observed. Seroconversion is defined as a rising of Legionella antibodies, dilution superior to 1/128 by indirect immunofluorescence. Nosocomial cases of Legionnaires' disease are defined in this study as the ones having an onset of symptoms more than 10 days after hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 3 years
  All cause mortality
Severity respiratory failure | 3 years
  Arterial pression of oxygen inferior to 600mmHg at diagnosis

SECONDARY OUTCOMES:
Age | One day
  Age at diagnosis
Sex | One day
  Sex
Charlson comorbidity index | One day
  This is a health tool that assesses the comorbidity risk associated to a series of conditions in order to offer medical specialists an informed decision making process in terms of specific screenings or medical procedures.The index accounts for the patient age and 16 different conditions, and ranges from 0 till 37.
Smoking status | One day
  Smoking (yes/no) at diagnosis
Nosocomial disease (yes/no) | One day
  Nosocomial cases of Legionnaires' disease are defined in this study as having an onset of symptoms more than 10 days after hospitalization.
C reactive protein | One day
  C reactive protein level at diagnosis
White blood cells | One day
  White blood cells level at diagnosis
Creatinine | One day
  Creatinine level at diagnosis
Urea | One day
  Urea level at diagnosis
Chest X Ray | One day
  Descriptive analysis of Chest X Ray findings at diagnosis
Method of diagnosis | One day
  Name of the method of diagnosis (urinary antigen, seroconversion, cultures).
Intensive care unit hospitalization | One day
  Intensive care unit hospitalization (yes/no)
Antibiotics | One day
  Name of antibiotics given
Antibiotic treatment duration | up to 40 days
  Antibiotic treatment duration

CONTACTS AND LOCATIONS:
Overall Officials: Marco Moretti, MD, Principal Investigator — CHU Brugmann
Locations (3):
- Belgium (3):
  - CHU Brugmann, Brussels
  - CHU St Pierre Hospital, Brussels
  - Universitair Zienkenhuis Brussel, Brussels

IPD SHARING:
Plan to Share IPD: No